CLINICAL TRIAL: NCT01381146
Title: Phase 1-2 Study of Victim Impact Group Modules for Jail Inmates
Brief Title: Victim Impact Modules for Jail Inmates
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from Phase II Study did not support "dismantling"
Sponsor: George Mason University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, June Tangney, Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA014694-12 (NIH); R01DA014694 (NIH)
Record Dates: First submitted 2011-06-17; First posted 2011-06-27 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Substance Abuse; HIV Risk; Shame; Guilt; Empathy; Criminogenic Thinking
Keywords: criminal behavior; substance abuse; HIV risk behavior; criminogenic thinking; shame; guilt; empathy; jail inmates; restorative justice; Crime
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impact of Crime Modules (Experimental): 5 session/1 week modules of a restorative justice inspired victim impact group intervention
  Interventions: Behavioral: Impact of Crime Modules
- TAU (Other): treatment as usual -- participants have access to all other jail programs and services
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Impact of Crime Modules — 5 session/1 week modules of a restorative justice inspired victim impact group intervention
  Arms: Impact of Crime Modules
Behavioral: TAU — have access to other jail programs and services
  Arms: TAU

SUMMARY:
The purpose of this study is to evaluate feasibility of modularized delivery of the Impact of Crime (IOC) group intervention with jail inmates, and obtain preliminary data on its effectiveness in reducing post-release recidivism, substance abuse, and HIV risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must be male
* Must be currently incarcerated jail inmate
* Must be sentenced
* Sentence must be short enough to serve out sentence at ADC
* Release date must follow projected final session of treatment
* Must speak, read, and write in English with sufficient proficiency to use workbook and participate in group sessions
* Must be assigned to the jail's "general population"

Exclusion Criteria:

* Actively psychotic
* Assigned "keep separate" from other group members

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Recidivism - Self report of arrests and undetected crimes | 3 months post-release up to 9 mos
Acceptability - number of participants who indicate the module was helpful and number who would recommend treatment to a friend | 1 week post-treatment up to 2 weeks
Number of inmates who complete the intervention | 5 sessions over a period of 1 week

SECONDARY OUTCOMES:
Self reported Substance use and dependence -Texas Christian University measure | 3 months post-release up to 9 mos
Self reported HIV risk behavior (sex and Intravenous Drug Use) Texas Christian University measure | 3 months post-release up to 9 mos
Changes in self-reported Shame-proneness from baseline | Changes from pre- to post-treatment up to 12 weeks
Changes in self-reported Shame-proneness from baseline | Changes from pre-treatment to 3 mos post-release up to 9 mos
Changes in self-reported Guilt-proneness from baseline | Changes from pretreatment to 3 months post-release up to 9 mos
Changes in self-reported Guilt-proneness from baseline | Changes from pretreatment to post-treatment up to 12 weeks
Changes in self-reported empathy from baseline | changes from pre- to post-treatment up to 12 weeks
Changes in self-reported empathy from baseline | changes from pre-treatment to 3 mos post-release up to 9 mos
Changes in self reported criminogenic thinking from baseline | changes from pre-treatment to post-treatment up to 12 weeks
Changes in self reported criminogenic thinking from baseline | changes from pre-treatment to 3 mos post-release up to 9 mos

CONTACTS AND LOCATIONS:
Overall Officials: June P Tangney, Ph.D., Principal Investigator — George Mason University
Locations (1):
- Fairfax County Adult Detention Center, Fairfax, Virginia, United States